CLINICAL TRIAL: NCT07193433
Title: Refinement, Pilot Implementation, and Testing of the Carer Support Needs Assessment Tool Intervention (CSNAT-I) in Hong Kong Palliative Care Settings
Brief Title: A Pilot Effectiveness and Implementation Trial of CSNAT-I in Hong Kong
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: United Christian Hospital (Other); Haven of Hope Hospital (Other)
Responsible Party: Principal Investigator, Dr CHENG Huilin, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 05; 20211161 (Other Grant/Funding Number: HMRF)
Record Dates: First submitted 2025-09-10; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Carers; Palliative Care; Needs Assessment; Supportive Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSNAT-I (Experimental)
  Interventions: Other: CSNAT-I
- Usual care (No Intervention): involve brief advice on stress management by healthcare providers on an informal basis

INTERVENTIONS:
Other: CSNAT-I — CSNAT-I will be conducted in five stages, including an introduction of the CSNAT, family caregivers' consideration of needs, prioritize needs, a shared care plan, and a shared review for effectiveness and subsequent actions .
  Arms: CSNAT-I

SUMMARY:
In this hybrid Type 1 effectiveness-implementation pilot randomized controlled trial, 60 caregivers will be randomized into either the CSNAT-I group or usual care. Preliminary effectiveness outcomes include caregiver burden, distress, and health-related quality of life. Preliminary implementation outcomes include feasibility, fidelity, appropriateness, acceptability, cost of the intervention, as well as barriers and facilitators to intervention implementation. Quantitative data will be analyzed using descriptive analysis and linear mixed effects model, while qualitative data using thematic analysis. The CSNAT-I is expected to be preliminarily effective in improving caregiver outcomes and implementable in Hong Kong palliative care context, which will serve as the foundation for a large trial before integration into daily practice.

ELIGIBILITY:
Inclusion Criteria

* adults ≥18 years old;
* family members taking a primary role in patient care at home as nominated by the palliative cancer patient;
* ability to communicate in Chinese.

Exclusion Criteria:

* paid caregivers;
* unable to complete the questionnaire due to mental impairment determined by physicians.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
Caregiver burden | From enrollment to the end of intervention at 4 weeks
  13-item Caregiver Strain Index (CSI), each item with 1 ("yes") or 0("no") responses. The total score ranges from 0 to 13 and a higher score represents greater caregiver burden.

SECONDARY OUTCOMES:
Caregiver distress | From enrollment to the end of intervention at 4 weeks
  The Depression, Anxiety, and Stress Scale (DASS), 4-point Likert scale ranging from 0('did not apply to me at all") to 3('applied to me very much'). The scale has 3 subscales, and the subscale score is obtained by summing up the item scores. A possible score range of 0 to 21 is each subscale. A higher score indicates greater depression, anxiety and stress.
Health-related quality of life | From enrollment to the end of intervention at 4 weeks
  Quality of Life in Life-Threatening Illness-Family Carer (QOLLTI-F), assesses seven dimensions, encompassing environment, patient condition, your own condition, your outlook, quality of care, relationships, and financial worries. The rating scale of each tool ranges from 0 to 10, and the total score is 160 respectively, with a higher total score indicating better QOL.
Reach | Through study completion, an average of 6 months
  eligibility rate, consent rate, participation rate, and reasons for non-participation will be used to measure reach of the intervention. All data will be collected from the study screening log.
Implementation | Through study completion, an average of 6 months.
  Fidelity, appropriateness and acceptability of the intervention, enablers and barriers to intervention implementation as well as the cost of the implementation. Fidelity of the intervention will be measured through the intervention delivery log. The appropriate and acceptability of the intervention, enablers and barriers to the intervention implementation will be collected using a self-designed questionnaire completed by participants. The cost of the implementation of the study will be calculated based on the time of interventionists for each intervention case multiplied by hourly salary determined by the hospital authority
Enablers and barriers to access, effectiveness, implementation, adoption, and maintenance | Up to 6 months
  We will explore enablers and barriers to access, effectiveness, implementation, adoption, and maintenance through meetings with hospital administration staff, health-related representatives and researchers before the completion of the study

IPD SHARING:
Plan to Share IPD: No